CLINICAL TRIAL: NCT04445792
Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics
Brief Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics (DCRI Coordinating Center)
Acronym: ADOPT PGx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00104948
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Depression; Acute Pain; Chronic Pain
Keywords: Pharmacogenetic; CYP2D6; CYP2C19
MeSH Terms: conditions — Depression; Acute Pain; Chronic Pain | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Immediate vs. delayed pharmacogenetic testing and genotype-guided pain or depression therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Acute Pain - Immediate PGx Testing (Experimental): Immediate genetic testing of CYP2D6 and clinical decisions support for pain management prescribing to the healthcare provider
  Interventions: Other: Pharmacogenetic testing; Other: Clinical decisions support
- Acute Pain - Delayed PGx Testing (Other): Delayed genetic testing of CYP2D6 and return of results after the conclusion of the 6-month follow-up period
  Interventions: Other: Pharmacogenetic testing
- Chronic Pain - Immediate PGx Testing (Experimental): Immediate genetic testing of CYP2D6 and clinical decisions support for pain management prescribing to the healthcare provider
  Interventions: Other: Pharmacogenetic testing; Other: Clinical decisions support
- Chronic Pain - Delayed PGx Testing (Other): Delayed genetic testing of CYP2D6 and return of results after the conclusion of the 6-month follow-up period
  Interventions: Other: Pharmacogenetic testing
- Depression - Immediate PGx Testing (Experimental): Immediate genetic testing of CYP2D6 and CYP2C19 and clinical decisions support for antidepressant prescribing to the healthcare provider
  Interventions: Other: Pharmacogenetic testing; Other: Clinical decisions support
- Depression - Delayed PGx Testing (Other): Delayed genetic testing of CYP2D6 and CYP2C19 and return of results after the conclusion of the 6-month follow-up period
  Interventions: Other: Pharmacogenetic testing

INTERVENTIONS:
Other: Pharmacogenetic testing — Genetic testing of CYP2D6 and CYP2C19
Other: Clinical decisions support — Prescribing recommendations to the provider based on the pharmacogenetic testing results
  Arms: Acute Pain - Immediate PGx Testing; Chronic Pain - Immediate PGx Testing; Depression - Immediate PGx Testing

SUMMARY:
This is a Master Protocol Screening record. This study is comprised of three separate pharmacogenetic trials grouped into a single protocol due to similarities in the intervention, the hypotheses, and the trial design. The three trials are the Acute Pain Trial, the Chronic Pain Trial, and the Depression Trial. Participants can enroll in only one of the three trials.

Each trial is listed individually on clinicaltrials.gov and includes "PRO00104948" within the Unique Protocol ID:

PRO00104948_A - Acute Pain Trial - NCT05966129

PRO00104948_B - Chronic Pain Trial - NCT05966142

PRO00104948_C - Depression Trial - NCT05966155

Acute Pain Trial: A prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided post-surgical opioid therapy (Intervention arm) or standard care and pharmacogenetic testing after 6 months (Control arm). The investigators will test the hypothesis that pharmacogenetic testing and genotype guided pain management therapy improves pain control after surgery in participants who's body processes some pain medicines slower than normal.

Chronic Pain Trial: A prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided opioid therapy (Intervention arm) or standard care with 6-month delayed pharmacogenetic testing (Control arm). The investigators will test the hypothesis that pharmacogenetic testing and genotype guided pain therapy improves pain control after surgery in participants who's body processes some pain medicines slower than normal.

Depression: A prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided anti-depressant therapy (Intervention arm) or standard care with 6-month delayed pharmacogenetic testing (Control arm). The investigators will test the hypothesis that pharmacogenetic testing and genotype-guided anti-depressant therapy will reduce depression symptoms in participants who's body processes some anti-depressants faster or slower than normal.

DETAILED DESCRIPTION:
Pain and depression are conditions that impact substantial proportions of the US population. Finding safe and effective drug therapies for both conditions is challenging. In the case of treatment for acute and chronic pain, the challenge is finding effective therapy while minimizing adverse effects or opioid addiction (and the ensuing consequences). For depression, there are few clinically relevant predictors of successful treatment leading to multiple trials of inadequate therapy for some patients. Both opioid and antidepressant prescriptions can be guided by pharmacogenetics (PGx) data based on existing guidelines from the Clinical Pharmacogenetics Implementation Consortium (CPIC).

This study is designed to evaluate the impact of pharmacogenetic testing and genotype-guided pain or anti-depressant therapy on pain control or depression symptoms in a pragmatic setting.

The rationale for examining a genotype-guided approach to acute and chronic pain management is based on the importance of CYP2D6 for the bioactivation of tramadol, codeine, and hydrocodone and data from a pilot study supporting improved pain control in intermediate and poor CYP2D6 metabolizers in the genotype-guided arm who are taking these drugs at baseline. Similarly, the rationale for examining a genotype-guided approach to depression medication therapy is based on the demonstrated role of CYP2D6 in the bio inactivation and CYP2C19 oxidation of select, commonly used SSRIs. Secondly, data from industry sponsored trials support the hypothesis of improved depression symptom control in a genotype-guided arm.

Study objectives:

Acute Pain Trial: Determine if a genotype-guided approach to acute post-surgical pain therapy leads to improved pain control compared to usual care, as defined by a decrease in the SIA score. Secondarily, The investigators will evaluate whether this approach leads to reduced use of DEA Schedule II opioids and reduced pain intensity.

Chronic Pain Trial: Determine if a genotype-guided approach to pain therapy in participants with at least 3 months of chronic pain leads to improved pain control compared to usual care.

Depression Trial: Determine if genotype-guided dosing or selection of antidepressants among participants with at least 3 months of depressive symptoms who require new or revised antidepressant therapy leads to improved control of depression, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Acute Pain

* Age ≥ 8 years
* English speaking or Spanish speaking
* Elective/planned surgery types with planned or anticipated to be treated with tramadol, hydrocodone, or codeine pain management at an enrolling site, which may include orthopedic surgeries (e.g. arthroplasty, spine, etc.), open abdominal surgery, or cardiothoracic surgery and others

Chronic Pain

* Age ≥ 18 years
* English speaking or Spanish speaking
* Seen at primary care clinics (such as, but not limited to, Internal Medicine, Family Medicine or Pediatrics) or patients seen in pain-relevant specialty clinics
* History of pain for at least the last 3 months
* Currently treated or being considered for treatment with tramadol, hydrocodone, or codeine to improve pain management

Depression

* Age ≥ 8 years
* English speaking or Spanish speaking
* Patients followed at psychiatry clinics or primary care clinics at an enrolling site (such as, but not limited to, Internal Medicine, Family Medicine, or Pediatrics)
* Documentation of depression and/or provider report of depression
* Evidence of depressive symptoms for at least 3 months based on patient interview or documentation in electronic health records
* Recent initiation of SSRI therapy, recent revised SSRI therapy, or anticipated need for revised or new SSRI therapy per health care provider

Exclusion Criteria

Trial-wide:

* Life expectancy less than 12 months
* Are too cognitively impaired to provide informed consent and/or complete study protocol
* Are institutionalized or too ill to participate (i.e. mental or nursing home facility or incarcerated)
* Have a history of allogeneic stem cell transplant or liver transplant
* People with prior clinical pharmacogenetic test results for genes relevant for the study in which they will enroll (CYP2D6 for the pain studies and CYP2D6 or CYP2C19 for depression) or already enrolled in an ADOPT PGx trial

Acute Pain

* Undergoing a laparoscopic surgery
* Receiving chronic opioid therapy, defined as use of opioids on most days for >3 months

Chronic Pain

* Plan to move out of the area within 6 months of enrollment
* Undergoing treatment for an active cancer diagnosis
* Currently taking daily opioids other than tramadol, codeine or hydrocodone

Depression

* Plan to move out of the area within 6 months of enrollment
* Have active psychosis or diagnosed psychotic disorders (schizophrenia, schizoaffective disorder, delusional disorder, psychotic depression, substance induced psychosis, schizophreniform disorder)
* Have dementia or other neurocognitive disorders due to any cause, such as Alzheimer's disease, vascular/subcortical, lewy body disease, frontotemporal lobar degeneration
* Have cognitive developmental delay and/or cognitive disability, including autism spectrum disorders (Note: ADHD is not an exclusion criteria)
* Has a seizure disorder
* Have bipolar disorder

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4284 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Chakraborty, Principal Investigator — Duke University
Locations (14):
- United States (14):
  - Nemours Children's Health System, Wilmington, Delaware
  - University of Florida - Gainesville, Gainesville, Florida
  - Nemours Children's Health System, Jacksonville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Nemours Children's Health System, Orlando, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Institute for Family Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Meharry Medical College, Nashville, Tennessee
  - Nashville General Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavallari LH, Cicali E, Wiisanen K, Fillingim RB, Chakraborty H, Myers RA, Blake KV, Asiyanbola B, Baye JF, Bronson WH, Cook KJ, Elwood EN, Gray CF, Gong Y, Hines L, Kannry J, Kucher N, Lynch S, Nguyen KA, Obeng AO, Pratt VM, Prieto HA, Ramos M, Sadeghpour A, Singh R, Rosenman M, Starostik P, Thomas CD, Tillman E, Dexter PR, Horowitz CR, Orlando LA, Peterson JF, Skaar TC, Van Driest SL, Volpi S, Voora D, Parvataneni HK, Johnson JA; IGNITE Pragmatic Trials Network. Implementing a pragmatic clinical trial to tailor opioids for acute pain on behalf of the IGNITE ADOPT PGx investigators. Clin Transl Sci. 2022 Oct;15(10):2479-2492. doi: 10.1111/cts.13376. Epub 2022 Aug 4. PMID 35899435
- [Background] Hines LJ, Wilke RA, Myers R, Mathews CA, Liu M, Baye JF, Petry N, Cicali EJ, Duong BQ, Elwood E, Hulvershorn L, Nguyen K, Ramos M, Sadeghpour A, Wu RR, Williamson L, Wiisanen K, Voora D, Singh R, Blake KV, Murrough JW, Volpi S, Ginsburg GS, Horowitz CR, Orlando L, Chakraborty H, Dexter P, Johnson JA, Skaar TC, Cavallari LH, Van Driest SL, Peterson JF; IGNITE Pragmatic Trials Network. Rationale and design for a pragmatic randomized trial to assess gene-based prescribing for SSRIs in the treatment of depression. Clin Transl Sci. 2024 Jun;17(6):e13822. doi: 10.1111/cts.13822. PMID 38860639
- [Background] Skaar TC, Myers RA, Fillingim RB, Callaghan JT, Cicali E, Eadon MT, Elwood EN, Ginsburg GS, Lynch S, Nguyen KA, Obeng AO, Park H, Pratt VM, Rosenman M, Sadeghpour A, Shuman S, Singh R, Tillman EM, Volpi S, Wiisanen K, Winterstein AG, Horowitz CR, Voora D, Orlando L, Chakraborty H, Van Driest S, Peterson JF, Cavallari LA, Johnson JA, Dexter PR; IGNITE Pragmatic Trials Network. Implementing a pragmatic clinical trial to tailor opioids for chronic pain on behalf of the IGNITE ADOPT PGx investigators. Clin Transl Sci. 2024 Aug;17(8):e70005. doi: 10.1111/cts.70005. PMID 39177194
- See also: Implementing a pragmatic clinical trial to tailor opioids for acute pain on behalf of the IGNITE ADOPT PGx investigators — https://pubmed.ncbi.nlm.nih.gov/35899435/
- See also: Rationale and design for a pragmatic randomized trial to assess gene-based prescribing for SSRIs in the treatment of depression — https://pubmed.ncbi.nlm.nih.gov/38860639/
- See also: Implementing a pragmatic clinical trial to tailor opioids for chronic pain on behalf of the IGNITE ADOPT PGx Investigators — https://pubmed.ncbi.nlm.nih.gov/39177194/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This record is for the overall master study protocol for the ADOPT PGx trial. The results for the individual trials are reported in separate records.
Pre-assignment Details: There were 4284 participants consented into the overall trial. Of the 4284, 174 consented participants were not randomized into the trial and were not assigned to a treatment arm. The remaining 4110 consented participants were randomized and assigned into the treatment arms. The 4110 randomized participants will be described moving forward.
Groups:
- Acute Pain, Chronic Pain, and Depression Trial Participants: Acute Pain Trial: A prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided post-surgical opioid therapy (Intervention arm) or standard care and pharmacogenetic testing after 6 months (Control arm).
  Chronic Pain Trial: A prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided opioid therapy (Intervention arm) or standard care with 6-month delayed pharmacogenetic testing (Control arm).
  Depression: A prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided anti-depressant therapy (Intervention arm) or standard care with 6-month delayed pharmacogenetic testing (Control arm).
Period: Overall Study
Arm/Group | Acute Pain, Chronic Pain, and Depression Trial Participants
Started | 4110
Completed | 3502
Not Completed | 608

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and will be in the ITT (intent to treat) population for the primary outcomes.
Arm/Group | Acute Pain, Chronic Pain, and Depression Trial Participants
Number analyzed (Participants) | 4110
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: <=18 years | 264
  Age, Categorical: 18 to 65 years | 2529
  Age, Categorical: >=65 years | 1317
  Age, Categorical: Unknown or Not Reported | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 2827
  Sex: Male | 1280
  Sex: Unknown or Not Reported | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 2782
  Gender: Male | 1276
  Gender: Transgender | 12
  Gender: Do not identify as female, male, or transgender | 28
  Gender: Prefer not to answer | 10
  Gender: Unknown | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 381
  Not Hispanic or Latino | 3679
  Unknown or Not Reported | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 29
  Asian | 71
  Native Hawaiian or Other Pacific Islander | 15
  Black or African American | 865
  White | 2671
  More than one race | 99
  Unknown or Not Reported | 360
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4110

OUTCOME MEASURES:

1. Primary Outcome: Number of Individuals Identified as Potential Participants Through EHR (Electronic Health Record)
Description: Potential participants identified for the Acute Pain, Chronic Pain, and Depression Trials through EHR.
Time Frame: Up to 3 years
Population: Individuals who were prescreened.
Measure: Count of Participants; unit: Participants
Groups:
- Individuals Identified as Potential Participants Through EHR: Potential participants for the Acute Pain, Chronic Pain, and Depression Trials.
Arm/Group | Individuals Identified as Potential Participants Through EHR
Number analyzed (Participants) | 77,451
Participants | 17,496

2. Primary Outcome: Number of Individuals Who Were Screened to the Acute Pain, Chronic Pain, and Depression Trials
Description: Individuals who were screened to be in the Acute Pain, Chronic Pain and Depression Trials.
Time Frame: Up to 3 years
Population: Individuals who were screened for the Acute Pain, Chronic Pain, and Depression Trials.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Pain, Chronic Pain, and Depression Trial Participants
Number analyzed (Participants) | 17,496
Participants | 4,285

3. Primary Outcome: Number of Participants Who Were Randomized to the Acute Pain, Chronic Pain, and Depression Trials
Description: Individuals who were randomized to be in the Acute Pain, Chronic Pain and Depression Trials.
Time Frame: Up to 3 years
Population: Participants who were consented to the Acute Pain, Chronic Pain, and Depression Trials.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Pain, Chronic Pain, and Depression Trial Participants
Number analyzed (Participants) | 4284
Participants | 4110

4. Secondary Outcome: Pain Interference as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS 43 subscale for pain interference assesses the extent to which participants experience interference with daily activities over the past 7 days using a 5-point Likert scale. The pain interference subscale provides a raw score ranging from 6 to 30. Raw scores are converted to T-scores using the PROMIS conversion tables, T-scores range from 41.1 to 76.3. Higher scores reflect greater pain interference.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 638 | 627 | 449 | 454 | 556 | 556
T-score | 51.0 (9.4) | 50.9 (9.6) | 62.4 (8.4) | 62.2 (8.6) | 51.7 (10.9) | 51.6 (11.2)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.7195, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.8054, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.861, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Physical Function as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS 43 subscale for physical functioning assesses a participants physical functioning over the past 7 days using a 5-point Likert scale. The physical functioning sub scale provides a raw score ranging from 6 to 30. Raw scores are converted to T-scores using the PROMIS conversion tables. T-scores range from 21.0 to 59.0. Higher T-scores reflect higher levels of physical functioning.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 642 | 627 | 447 | 455 | 557 | 556
T-score | 44.9 (9.7) | 45.3 (9.6) | 36.0 (7.5) | 36.2 (7.5) | 47.2 (9.7) | 46.8 (10.3)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.4385, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.7185, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.431, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Sleep Disturbance as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS 43 subscale for sleep disturbance assesses the extent to which participants experience sleep disturbance related symptoms sleep over the past 7 days using a 5-point Likert scale. The sleep disturbance subscale provides a raw score ranging from 6 to 30. Raw scores are converted to T-scores using the PROMNIS conversion tables, ranging from 31.7 to 76.1. Higher scores reflect higher levels of sleep disturbance.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 642 | 630 | 448 | 456 | 556 | 556
T-score | 48.5 (9.5) | 48.5 (9.5) | 55.3 (9.5) | 54.6 (9.6) | 53.8 (8.9) | 55.0 (8.8)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.9222, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.1918, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0119, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Ability to Participant in Social Roles and Activities as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS 43 subscale for ability to participate in social roles and activities assesses the extent to which participants are able to participant in different social roles and activities over the past 7 days using a 5-point Likert scale. The ability to participant in social roles and activities subscale provides a raw score ranging from 6 to 30. Raw scores are converted to T-scores using the PROMIS conversion tables, T-scores range from 26.7 to 65.0 with higher values corresponding to a higher ability to participant in social roles and activities.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 642 | 630 | 448 | 454 | 557 | 556
T-score | 53.4 (10.3) | 53.5 (10.3) | 44.2 (9.5) | 44.9 (9.8) | 49.4 (10.0) | 48.3 (10.3)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.6971, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.2309, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0441, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Fatigue as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS 43 subscale for fatigue assesses the extent to which participants experience fatigue-related symptoms over the past 7 days using a 5-point Likert scale. The fatigue subscale provides a raw score ranging from 6 to 30. Raw scores are converted to T-scores using the PROMIS conversion tables, T-scores range from 33.4 to 76.8. Higher T-scores reflect greater fatigue symptoms.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 640 | 623 | 448 | 456 | 557 | 556
T-score | 46.7 (10.2) | 46.6 (10.3) | 56.0 (10.8) | 54.7 (10.7) | 55.4 (9.8) | 57.0 (10.7)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.7988, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.0483, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0104, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Anxiety as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS subscale for anxiety assesses the extent to which participants experience anxiety symptoms over the past 7 days using a 5-point Likert scale. The anxiety subscale provides a raw score, ranging from 6 to 30. Raw scores are converted to T-scores using the PROMIS conversion tables, T-scores range from 33.4 to 76.8. Higher T-scores reflect greater anxiety.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 641 | 624 | 449 | 456 | 556 | 556
T-score | 45.5 (9.0) | 45.2 (9.0) | 52.7 (11.2) | 51.9 (11.2) | 57.5 (9.3) | 58.4 (9.9)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.521, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.2348, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0517, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Depression as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 6-item PROMIS 43 subscale for depression assesses the extent to which participants experience depressive symptoms over the past 7 days using a 5-point Likert scale. The depression subscale provides a raw sore ranging from 6 to 30. Raw scores are converted to T-scores using the PROMIS conversion tables, T-scores range from 38.4 to 80.3. Higher T-scores reflect greater depression.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 639 | 626 | 449 | 456 | 557 | 556
T-score | 44.0 (8.2) | 43.7 (7.9) | 51.2 (10.5) | 49.7 (10.6) | 55.0 (9.6) | 56.6 (9.9)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.6835, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.0205, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0036, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Overall Wellbeing as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: Overall wellbeing is the sum of the PROMIS 43 subdomain T-scores, with physical function and ability to participate in social roles scores reversed such that higher values within each subscale correspond with poorer health. Overall wellbeing ranges from 259.7 to 541.2, higher scores correspond to worse wellbeing.
Time Frame: 6 months
Population: Randomized population with completed 6 month survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 634 | 613 | 444 | 451 | 555 | 556
score on a scale | 337.4 (51.3) | 336.2 (51.2) | 397.6 (50.5) | 392.1 (50.7) | 376.8 (51.8) | 383.6 (53.5)
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p = 0.5878, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.1051, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0292, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Number of Participants With Pharmacogenetic Drug-Gene Concordance
Description: Concordance between PGx phenotypes and opioid (Acute Pain and Chronic Pain) and SSRI (Depression) medications.
Time Frame: 10 days for Acute Pain; 3 months for Chronic Pain and Depression
Population: Randomized population with completed 6 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Pain - Immediate PGx Testing | Acute Pain - Delayed PGx Testing | Chronic Pain - Immediate PGx Testing | Chronic Pain - Delayed PGx Testing | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Number analyzed (Participants) | 716 | 699 | 469 | 466 | 656 | 656
Participants | 642 | 548 | 371 | 362 | 609 | 579
Statistical Analysis 1: Comparison: Acute Pain - Immediate PGx Testing vs Acute Pain - Delayed PGx Testing; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Chronic Pain - Immediate PGx Testing vs Chronic Pain - Delayed PGx Testing; Test type: Superiority; p = 0.5973, Chi-squared
Statistical Analysis 3: Comparison: Depression - Immediate PGx Testing vs Depression - Delayed PGx Testing; Test type: Superiority; p = 0.0046, Chi-squared

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Description: Per the study protocol, only Adverse Device Effect (ADE) events suspected to be related to the specimen collection, laboratory assay genotyping results, and phenoconversion recommendations from the Best Practice Alerts (BPAs)/Consult notes were reported to the IRB. Reportable ADEs or unanticipated Adverse Device Effect (UADEs) events including unanticipated study related deaths will be collected in the study database per IRB reporting policies. Medication side effects were not included as AEs.
Groups:
- Immediate Pharmacogenetics (PGx) Guided Therapy: Acute Pain Trial: Immediate pharmacogenetic testing and genotype-guided post-surgical opioid therapy (Intervention arm).
  Chronic Pain Trial: Immediate pharmacogenetic testing and genotype-guided opioid therapy (Intervention arm).
  Depression: Immediate pharmacogenetic testing and genotype-guided anti-depressant therapy (Intervention arm).
- Delayed Pharmacogenetics (PGx) Testing: Acute Pain Trial: Standard care and pharmacogenetic testing after 6 months (Control arm).
  Chronic Pain Trial: Standard care with 6-month delayed pharmacogenetic testing (Control arm).
  Depression: Standard care with 6-month delayed pharmacogenetic testing (Control arm).
Arm/Group | Immediate Pharmacogenetics (PGx) Guided Therapy | Delayed Pharmacogenetics (PGx) Testing
All-Cause Mortality (participants affected / at risk) | 5/2055 | 7/2055
Serious Adverse Events (participants affected / at risk) | 0/2550 | 0/2550
Other Adverse Events (participants affected / at risk) | 1/2550 | 0/2550
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Pharmacogenetics (PGx) Guided Therapy (N=2550) | Delayed Pharmacogenetics (PGx) Testing (N=2550)
Panic Attack due to sample blood draw (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04445792/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT04445792/ICF_000.pdf